CLINICAL TRIAL: NCT01124214
Title: In Vivo Endomicroscopy (EM) for Improved Diagnosis of Barrett's Esophagus (BE) and Associated Neoplasia: A Multicenter Randomized Controlled Trial of Diagnostic Yield and Clinical Impact
Brief Title: Confocal Endomicroscopy for Improved Diagnosis of Barrett's Esophagus and Early Esophageal Cancer(CEBE Study)
Acronym: CEBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other); Pentax Medical Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NA_00025471
Record Dates: First submitted 2010-05-13; First posted 2010-05-17 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Barrett's Esophagus, Esophageal Intraepithelial Neoplasia
Keywords: Barrett's; BE; esophageal cancer; esophageal dysplasia
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms | interventions — Eukaryotic Initiation Factor-2B; Microscopy, Confocal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Resolution endoscopy (HRE) (No Intervention): Standard of care, high resolution endoscopy surveillance/ evaluation of BE and or IEN
- Endomicroscopy (EM) (Active Comparator): Standard of care, high resolution endoscopy surveillance/ evaluation of BE and or IEN and endomicroscopy esophageal evaluation
  Interventions: Procedure: endomicroscopy

INTERVENTIONS:
Procedure: endomicroscopy — endomicroscopy scope lens has capability to optically evaluate mucosa/submucosa as a microscope
  Other Names: Confocal Laser Microscopy (CLE), EM, confocal microscopy
  Arms: Endomicroscopy (EM)

SUMMARY:
Endomicroscopy (EM) can improve the diagnosis Barrett's esophagus (BE) and some early esophageal cancers (Intra Epithelial Neoplasia (IEN)). EM provides optical biopsies comparable to standard histology. Specifically, EM allows targeted biopsy rather than random mucosal biopsy during routine endoscopic surveillance of BE or evaluation EIN, which will improve the diagnostic yield of mucosal samples for BE IEN. Furthermore, when combined with high resolution endoscopy, EM may improve the overall in vivo detection of IEN in lesions as well as flat mucosa.

EM will provide accurate place and size of IEN which will impact the physician's decision to biopsy or perform endoscopic mucosal resection (EMR). This could potentially minimize the number of unnecessary biopsies and as well as enable the physician to perform EMR at the time of the initial examination, rather than delaying endoscopic treatment after the pathology is available. This study is important because it will validate single center studies supporting the routine use of EM for screening and surveillance of BE.

DETAILED DESCRIPTION:
The central hypothesis is that endomicroscopy (EM) can improve the efficiency of the endoscopic diagnosis of Barrett's esophagus (BE) and associated Intraepithelial neoplasia(IEN), providing in-vivo optical biopsies comparable to standard histology. Specifically, EM will enable targeted biopsy rather than random mucosal biopsy during routine endoscopic surveillance of BE or endoscopic evaluation of patients with suspected or proven unlocalized IEN, which will improve the diagnostic yield of mucosal samples for BE IEN. Furthermore, when combined with high resolution endoscopy, EM may improve the overall in vivo detection of IEN in lesions as well as flat mucosa.

The investigators also hypothesize that EM will provide additional accurate information regarding the presence of IEN that will impact upon the physician's decision to obtain a mucosal biopsy or perform endoscopic mucosal resection (EMR). This could potentially minimize the number of unnecessary biopsies and as well as enable the physician to perform EMR at the time of the initial examination, rather than delaying endoscopic treatment to another procedure after the pathology from the mucosal biopsies are available. This study is important because it will validate single center studies supporting the routine use of EM for screening and surveillance of BE.

ELIGIBILITY:
Inclusion Criteria:

* Surveillance of Barrett's esophagus or suspected or known BE associated neoplasia

Exclusion Criteria:

* Allergy or prior reaction to the fluorescent contrast agent fluorescein sodium
* Unable to give informed consent.
* Pregnant or breastfeeding women
* Known advanced adenocarcinoma in the esophagus
* Dysplastic or suspected malignant esophageal lesion 0 BE lesions 2 cm or more in size with Paris classification of 0-Ip (polypoid), 0-Is (protruding sessile), 0-IIa (flat elevated), or 0-IIb (flat)
* Lesions of any size with Paris 0-IIc (superficial shallow depressed) or 0-III (excavated)
* Acute gastrointestinal bleeding
* Coagulopathy defined by Partial Thromboplastin Time (PTT) > 50 sec, or International Normalized Ratio (INR) > 2.0, platelets < 40,000, or on chronic anticoagulation
* Inability to tolerate sedated upper endoscopy due to cardio-pulmonary instability or other contraindication to endoscopy.
* History of a severe allergic reaction (anaphylaxis)
* Known, untreated esophageal strictures, prior partial esophageal resection, or altered anatomy preventing passage of the endomicroscope

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
compare diagnostic yield | 1 year
  Compare the diagnostic yield (defined as the proportion of mucosal biopsy samples with neoplasia) of HRE plus EM with directed biopsy (HRE-EM-DB) over HRE with directed biopsy of all mucosal lesions followed by random biopsy (HRE-DB-RB) to diagnose BE in flat mucosa and mucosal lesions
  The mean diagnostic yield for IEN will be calculated (number of mucosal biopsies and EMR specimens with High Grade Dysplasia (HGD) or Carcinoma (CA) divided by total number of mucosal biopsies obtained) by group and compared, using a chi square or Fisher's exact test for independent groups, depending on the distribution of the data.

SECONDARY OUTCOMES:
assess clinical impact of EM | 1 year
  To prospectively assess the potential clinical impact of EM on the diagnosis and endoscopic surveillance of BE by determining if EM alters the decision to biopsy or EMR and change the total of biopsies per procedure.
compare the specificity and sensitivity of HRE with EM | 1 year
  To compare the performance (sensitivity and specificity) characteristics of HRE-EM-DB with HRE-RB for prediction of BE/IEN using the pathologic diagnosis of mucosal biopsies the as the reference standard.

CONTACTS AND LOCATIONS:
Overall Officials: Marcia I Canto, MD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mount Sinai School of Medicine, New York, New York
  - University of Pennsylvania Medical Institution, Philadelphia, Pennsylvania
- Johannes Gutenberg - University of Mainz, Mainz, Germany

REFERENCES:
- [Background] Canto MI, Anandasabapathy S, Brugge W, Falk GW, Dunbar KB, Zhang Z, Woods K, Almario JA, Schell U, Goldblum J, Maitra A, Montgomery E, Kiesslich R; Confocal Endomicroscopy for Barrett's Esophagus or Confocal Endomicroscopy for Barrett's Esophagus (CEBE) Trial Group. In vivo endomicroscopy improves detection of Barrett's esophagus-related neoplasia: a multicenter international randomized controlled trial (with video). Gastrointest Endosc. 2014 Feb;79(2):211-21. doi: 10.1016/j.gie.2013.09.020. Epub 2013 Nov 9. PMID 24219822
- See also: Johns Hopkins GI website, Barrett's esophagus section — https://www.ncbi.nlm.nih.gov/pubmed/?term=In+vivo+endomicroscopy+improves+detection+of+Barrett%E2%80%99s+esophagus%E2%80%93related+neoplasia%3A+a+multicenter+international+randomized+controlled+trial